CLINICAL TRIAL: NCT00421993
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Study to Demonstrate the Efficacy and Safety of Adapalene/Benzoyl Peroxide Topical Gel Compared With Adapalene Topical Gel, 0.1%; Benzoyl Peroxide Topical Gel, 2.5% and Topical Gel Vehicle in Subjects With Acne Vulgaris
Brief Title: A Study to Demonstrate the Efficacy and Safety of Adapalene/Benzoyl Peroxide Topical Gel in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Michael Graeber, MD, Head of US Development, Galderma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18088
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2009-03-11 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2009-10

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Adapalene; Benzoyl Peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): Adapalene/Benzoyl Peroxide Topical Gel
  Interventions: Drug: Adapalene/Benzoyl Peroxide
- 2 (Active Comparator): Adapalene Topical Gel
  Interventions: Drug: Adapalene
- 3 (Active Comparator): Benzoyl Peroxide Topical Gel
  Interventions: Drug: Benzoyl Peroxide
- 4 (Placebo Comparator): Topical Gel Vehicle
  Interventions: Drug: Topical Gel Vehicle

INTERVENTIONS:
Drug: Adapalene/Benzoyl Peroxide — Topical Gel, One application daily in the evening for 12 weeks
  Arms: 1
Drug: Adapalene — Topical Gel,One application daily in the evening for 12 weeks
  Arms: 2
Drug: Benzoyl Peroxide — Topical Gel, one application daily in the evening for 12 weeks
  Arms: 3
Drug: Topical Gel Vehicle — Topical Gel Vehicle,one application daily in the evening for 12 weeks
  Arms: 4

SUMMARY:
This is a multi-center, randomized, double-blind, parallel group study with 12 weeks of treatment of acne vulgaris. Efficacy and safety evaluations will be performed at Screening (safety only), Baseline and Weeks 1, 2, 4, 8 and 12. All Investigator's Global Assessment evaluators and lesion counters must be trained and approved by Galderma. The evaluator of a subject should remain the same during the study.

The primary objective is to demonstrate the superiority in efficacy and assess safety of Adapalene/Benzoyl Peroxide Topical Gel (Adapalene/Benzoyl Peroxide Gel) versus Adapalene Topical Gel, 0.1% (Adapalene Monad); Benzoyl Peroxide Topical Gel, 2.5% (Benzoyl Peroxide Monad) and Topical Gel Vehicle (Gel Vehicle) in the treatment of acne vulgaris for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acne vulgaris with facial involvement.
* A minimum of 20 but not more than 50 Inflammatory lesions
* A minimum of 30 but not more than 100 Noninflammatory lesions
* A score of 3 (Moderate) on the Investigator's Global Assessment Scale.

Exclusion Criteria:

* More than one acne nodule or any acne cyst.
* Acne conglobata, acne fulminans, secondary acne, or severe acne.
* Known previous participation in an Adapalene/Benzoyl Peroxide Topical Gel Trial.
* Underlying diseases that require the use of interfering topical or systemic therapy.
* Use of prohibited medications prior to the study unless appropriate washout period is documented
* Use of hormonal contraceptives solely for control of acne

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1670 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (62):
- United States (33):
  - Medical Affliated Research Center, Huntsville, Alabama
  - Dermatology Research of Arkansas, Little Rock, Arkansas
  - Associates in research, Inc., Fresno, California
  - University of California, Irvine, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Marcia J. Glenn, MD and Associates, Dermatology & Laser center, Inc, Marina del Rey, California
  - Affiliated Research Institute, San Diego, California
  - University at San Francisco Medical Center, San Francisco, California
  - Radiant Research, Santa Rosa, California
  - Dr Weintraub James, Simi Valley, California
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Visions Clinical Research, West Palm Beach, Florida
  - Atlanta Dermatology and Vein Research Center, Alpharetta, Georgia
  - SKINQRI, Lincolnshire, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Hamzavi Dermatology, Port Huron, Michigan
  - Somerset Skin Clinic, Troy, Michigan
  - James Del Rosso, DO - Office of Dr. James Del Russo, Henderson, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Skin Specialty Group, New York, New York
  - Derm Research Center of NY, Inc., Stony Brook, New York
  - Zoe Draelos, High Point, North Carolina
  - OU Health Sciences Center - Dept. of Dermatology, Oklahoma City, Oklahoma
  - Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Radiant Research, Anderson, South Carolina
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - UTSW Medical Center at Dallas, Dallas, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Tanner Clinic, Layton, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
- Canada (15):
  - The Dermatology Centre, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Derm Research @ 888 Inc., Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Dermadvances Research, Winnipeg, Manitoba
  - Nexus clinical research, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research, St. John's, Newfoundland and Labrador
  - Ultranova Skin care, Barrie, Ontario
  - Lynderm Research inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
  - Innovaderm Research Laval Inc., Laval, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
- Germany (8):
  - Licca Clinical Research Institute, Augsburg
  - Henrik Pres, Berlin
  - Meike Schroeder, Berlin
  - Beatrice Gerlach, Dresden
  - Kloverkorn, Windfried, Gilching
  - Otto-Von-Guericke-Universitat Magdeburg, Magdeburg
  - Michael Sebastian, Mahlow
  - Thomas Dirschka, Wuppertal
- Hungary (3):
  - Outpatient Dermatology Department DUH, Budapest
  - Margit Simola, Budapest
  - Outpatient Dermatilogy Department XIX District, Budapest
- Poland (3):
  - Waldemar Placek, Bydgoszcz
  - DERMED Specjalistyczne Gabinety Lekarskie, Lodz
  - Wojceiech Silny, Poznan

REFERENCES:
- [Background] Leyden JJ. A review of the use of combination therapies for the treatment of acne vulgaris. J Am Acad Dermatol. 2003 Sep;49(3 Suppl):S200-10. doi: 10.1067/s0190-9622(03)01154-x. PMID 12963896
- See also: Related Info — http://www.galderma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: First Subject Enrolled October 2006, Last Subject Enrolled July 2007.
  Types of locations: Dermatology Clinics, Dermatology Research Centers.
Pre-assignment Details: The specified washout period up to Baseline for TOPICAL facial treatments was 1 week (light therapy/exfoliation/blackhead removal) or 2 weeks (anti-inflammatory drugs/salicylic acid/steroids/antibiotics/laser) and for SYSTEMIC medications was 2 weeks (anti-inflammatory drugs), 4 Weeks (steroids/antibiotics), or 6 months (anti-acne/contraceptives).
Groups:
- Adapalene/Benzoyl Peroxide Gel: Adapalene/Benzoyl Peroxide Topical Gel
- Adapalene Gel: Adapalene Topical Gel
- Benzoyl Peroxide Gel: Benzoyl Peroxide Topical Gel
- Gel Vehicle: Topical Gel Vehicle
Period: Overall Study
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Started | 419 | 418 | 415 | 418
Completed | 366 | 369 | 363 | 361
Not Completed | 53 | 49 | 52 | 57
Not completed — Withdrawal by Subject | 22 | 23 | 23 | 24
Not completed — Lost to Follow-up | 18 | 19 | 22 | 20
Not completed — Adverse Event | 11 | 1 | 6 | 4
Not completed — Protocol Violation | 2 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 3 | 0 | 5
Not completed — Pregnancy | 0 | 1 | 1 | 2
Not completed — Subject transportation issues | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle | Total
Number analyzed (Participants) | 419 | 418 | 415 | 418 | 1670
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (6.7) | 18.5 (6.3) | 18.9 (6.96) | 19.2 (7.23) | 19 (6.81)
Age, Customized [Number; unit: participants]
  12-17 years | 233 | 241 | 244 | 243 | 961
  Between 18 and 64 years | 186 | 177 | 171 | 175 | 709
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 229 | 230 | 244 | 939
  Male | 183 | 189 | 185 | 174 | 731
Region of Enrollment [Number; unit: participants]
  United States | 185 | 185 | 179 | 185 | 734
  Canada | 102 | 100 | 100 | 101 | 403
  Europe | 132 | 133 | 136 | 132 | 533

OUTCOME MEASURES:

1. Primary Outcome: Success Rate on the Investigator's Global Assessment
Description: Percentage of subjects rated "Clear" and "Almost Clear" on 5-point scale (0=clear; 4=severe)
Time Frame: at week 12
Population: Intention to treat (ITT), last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Percentage of participants | 37.9 | 21.8 | 26.7 | 17.9

2. Primary Outcome: Changes in Inflammatory Lesion Counts
Description: Changes in Inflammatory Lesion Counts equals Week 12 Inflammatory Lesion Counts minus Baseline Inflammatory Lesion Counts
Time Frame: from Baseline to week 12
Population: ITT, LOCF
Measure: Median (Full Range); unit: Lesion count
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Lesion count | -18 [-49 to 50] | -15 [-49 to 50] | -16 [-63 to 38] | -12 [-47 to 95]

3. Primary Outcome: Changes in Noninflammatory Lesion Counts
Description: Change in Noninflammatory Lesion Counts equals Week 12 Noninflammatory Lesion Count minus Baseline Noninflammatory Lesion Count
Time Frame: from Baseline to week 12
Population: ITT, LOCF
Measure: Median (Full Range); unit: Lesion count
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Lesion count | -28 [-93 to 108] | -24 [-96 to 44] | -23 [-87 to 61] | -18 [-82 to 69]

4. Secondary Outcome: Percent Change in Inflammatory Lesion Counts
Description: Percent Changes in Inflammatory Lesion Counts equals (Week 12 count minus Baseline count) divided by Baseline count multiplied by 100
Time Frame: at week 12
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Percent change | -61.7 (33.9) | -50.1 (39.4) | -52.2 (39.4) | -40.8 (41.1)

5. Secondary Outcome: Percent Change in Noniflammatory Lesion Counts
Description: Percent Changes in Noninflammatory Lesion Counts equals (Week 12 count minus Baseline count) divided by Baseline count multiplied by 100
Time Frame: at week 12
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Percent change | -55.6 (35.3) | -46.0 (33.7) | -44.1 (37.3) | -32.3 (39.5)

6. Secondary Outcome: Percent Change in Total Lesion Counts
Description: Percent Changes in Total Lesion Counts equals (Week 12 count minus Baseline count) divided by Baseline count multiplied by 100
Time Frame: at week 12
Population: ITT, LOCF
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Number analyzed (Participants) | 419 | 418 | 415 | 418
Percent change | -57.7 (31.9) | -47.5 (31.3) | -47.2 (32.7) | -35.2 (36)

ADVERSE EVENTS:
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel | Benzoyl Peroxide Gel | Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 3/419 | 1/418 | 1/415 | 2/418
Other Adverse Events (participants affected / at risk) | 90/419 | 60/418 | 35/415 | 22/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/Benzoyl Peroxide Gel (N=419) | Adapalene Gel (N=418) | Benzoyl Peroxide Gel (N=415) | Gel Vehicle (N=418)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/Benzoyl Peroxide Gel (N=419) | Adapalene Gel (N=418) | Benzoyl Peroxide Gel (N=415) | Gel Vehicle (N=418)
Dry Skin (Skin and subcutaneous tissue disorders) | 90 (93) | 60 (61) | 35 (37) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the expiration of twenty-four (24) months after the completion of the Study, Investigator shall have the right to publish the results of the Study; provided, however that Sponsor shall have the right to review any proposed publication generated from the Study prior to publication or presentation. The Sponsor shall have the absolute right to refuse the publication altogether, to delay it or to amend its contents as it deems fit.